CLINICAL TRIAL: NCT03829293
Title: High-Flow Nasal Oxygenation Versus Standard Oxygenation in Gastrointestinal Endoscopy With Sedation. A Prospective Multicenter Randomized Study
Brief Title: High-Flow Nasal Oxygenation Versus Standard Oxygenation in Gastrointestinal Endoscopy With Sedation.
Acronym: ODEPHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRO-2019-01
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Gastrointestinal Endoscopy; Sedation
Keywords: High-flow nasal cannula oxygenation; gastrointestinal endoscopy; upper gasatrointestinal endoscopy; colonoscopy; sedation; hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal cannula oxygenation group (Experimental): Participants in the experimental group will receive high-flow nasal oxygen therapy (HFNO) during gastrointestinal endoscopy under sedation (with a flow at 70L/min and oxygen inspired fraction (FiO2) 50%) through a dedicated system, the THRIVETM (Fisher&Paykel, New-Zealand)
  Interventions: Device: High-flow nasal cannula oxygenation group
- Standard Oxygenation (No Intervention): Participants in the current standard of care will receive standard oxygenation by nasal prongs (with a flow at 6L/min) or naropharyngeal catheter (with a flow at 5L/min) or standard face mask (with a flow at 6L/min)

INTERVENTIONS:
Device: High-flow nasal cannula oxygenation group — usual care + High-flow nasal oxygenation (HFNO) therapy during GI endoscopy under sedation (with a flow at 70L/min and FiO2 50%) through a dedicated system, the THRIVETM (Fisher&Paykel, New-Zealand)
  Arms: High-flow nasal cannula oxygenation group

SUMMARY:
This study is a randomized controlled trial comparing high-flow nasal oxygen therapy (HFNO) versus standard oxygen therapy (nasal prongs, nasopharyngeal catheter or standard face mask) during gastrointestinal (GI) endoscopy with sedation to reduce the incidence of hypoxia.

DETAILED DESCRIPTION:
Hypoxemia is the most common complication during a gastrointestinal endoscopy with sedation. Oxygenation is usually applied during the procedure to prevent the occurrence of desaturation. Conventional oxygen is typically administered by conventional nasal cannula, by nasopharyngeal catheter or by a facemask with mild flow of oxygen. The flow of standard oxygen is limited to 15L/min.

High-flow nasal cannula oxygenation is a new method of humidified and heated oxygenation with a higher flow rates (up to 70L/min).

The primary outcome will be the incidence of hypoxia defined by pulsed saturation with oxygen (SpO2) ≤92%. The investigator's hypothesis is that high-flow nasal oxygen therapy will decrease the frequency of hypoxemia during gastrointestinal endoscopy under sedation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Having GI endoscopy expected under sedation
* At risk of hypoxia defined by (one of the item): an underlying cardiac disease ; an underlying respiratory disease ; age greater than or equal to 60 years ; ASA II, III or ASA IV ; with an body mass index greater or equal to 30 (kg/m²); with sleep apnea syndrome diagnosed or suspected with a STOP-BANG score ≥ 3

Exclusion Criteria:

* Age below 18
* Emergency GI endoscopy
* Need of intubation for the procedure
* Patient with chronic oxygen treatment
* Patients with tracheostomy
* Pregnancy, breastfeeding
* Not affiliated to French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoxia | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  SpO2 ≤ 92%

SECONDARY OUTCOMES:
Incidence of hypoxia in the recovery room | Length of stay in the recovery room, an expected average of 2 hours
  SpO2 ≤ 92%
Incidence of apnea during the procedure | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  Breath rate ≤6/min
Incidence of hypoxia with SpO2 ≤ 90% | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  SpO2 ≤ 90%
Incidence of severe hypoxia | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  SpO2 ≤ 85%
Prolonged hypoxia during the procedure | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  SpO2 ≤ 92% for ≥60 s
Severe hypoxia during the procedure | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  SpO2 ≤ 90% and SpO2 ≤85%
Modification of oxygenation during the procedure | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  Increase of oxygen flow in conventional group or FiO2 in the interventional group to maintain an adequate oxygenation
The need of intervention by the anesthesia team | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  Need of airway manipulation, use of noninvasive ventilation or mechanical invasive ventilation
Temporal course of SpO2 | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  Absolute changes in SpO2
Temporal course of respiratory rate | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  Absolute changes in respiratory rate, in cycles/minutes
Temporal course of heart rate | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  Absolute changes in heart rate, in bpm
Temporal course of arterial blood pressure | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  Absolute changes arterial blood pressure, in mmHg
Incidence of bradycardia | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  Heart rate < 50 bpm
Incidence of need for mechanical respiratory support | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  noninvasive ventilation, or ventilation through a laryngeal mask, or tracheal intubation
Failure of the endoscopic procedure | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  Number of patients in whom the endoscopic procedure has to be stopped and postponed
Duration of the endoscopic procedure | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  From insertion of the fiberoptic endoscope to its withdrawal, in minutes
Duration of sedation | Duration of GI endoscopy procedure under sedation, an expected average of 2 hours
  From anaesthesia induction to the awakening of the patient, in minutes
Length of stay in the recovery room | Length of stay in the recovery room, an expected average of 2 hours
  From admission at to discharge from the recovery room, in minutes
Need of hospitalisation | 24 hours
  percentage of ambulatory patients who needed to be hospitalised after the procedure
Serious adverse event rate | 24 hours
  Percentage of patients experiencing at least one serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh NAY, Dr, Study Director — CHR Orléans; Willy-Serge MFAM, Dr, Principal Investigator — CHR Orléans; Olivier BAERT, Dr, Principal Investigator — Pôle Santé Oréliance; Adrien AUVET, Dr, Principal Investigator — CH de Dax; Francis REMERAND, Dr, Principal Investigator — CHU de Tours - hôpital Trousseau
Locations (3):
- France (3):
  - Hospital Center of DAX, Dax
  - Pole santé ORELIANCE, Orléans
  - Orleans Hospital Center, Orléans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Qadeer MA, Lopez AR, Dumot JA, Vargo JJ. Hypoxemia during moderate sedation for gastrointestinal endoscopy: causes and associations. Digestion. 2011;84(1):37-45. doi: 10.1159/000321621. Epub 2011 Feb 8. PMID 21304242
- [Result] Qadeer MA, Rocio Lopez A, Dumot JA, Vargo JJ. Risk factors for hypoxemia during ambulatory gastrointestinal endoscopy in ASA I-II patients. Dig Dis Sci. 2009 May;54(5):1035-40. doi: 10.1007/s10620-008-0452-2. Epub 2008 Nov 12. PMID 19003534
- [Result] Cohen LB, Wecsler JS, Gaetano JN, Benson AA, Miller KM, Durkalski V, Aisenberg J. Endoscopic sedation in the United States: results from a nationwide survey. Am J Gastroenterol. 2006 May;101(5):967-74. doi: 10.1111/j.1572-0241.2006.00500.x. PMID 16573781
- [Result] Griffin SM, Chung SC, Leung JW, Li AK. Effect of intranasal oxygen on hypoxia and tachycardia during endoscopic cholangiopancreatography. BMJ. 1990 Jan 13;300(6717):83-4. doi: 10.1136/bmj.300.6717.83. No abstract available. PMID 2105779
- [Result] Woods A, Sanowski RA, Wadas DD, Manne RK, Friess SW. Eradication of diminutive polyps: a prospective evaluation of bipolar coagulation versus conventional biopsy removal. Gastrointest Endosc. 1989 Nov-Dec;35(6):536-40. doi: 10.1016/s0016-5107(89)72906-0. PMID 2689263
- [Derived] Nay MA, Fromont L, Eugene A, Marcueyz JL, Mfam WS, Baert O, Remerand F, Ravry C, Auvet A, Boulain T. High-flow nasal oxygenation or standard oxygenation for gastrointestinal endoscopy with sedation in patients at risk of hypoxaemia: a multicentre randomised controlled trial (ODEPHI trial). Br J Anaesth. 2021 Jul;127(1):133-142. doi: 10.1016/j.bja.2021.03.020. Epub 2021 Apr 28. PMID 33933271
- [Derived] Eugene A, Fromont L, Auvet A, Baert O, Mfam WS, Remerand F, Boulain T, Nay MA. High-flow nasal oxygenation versus standard oxygenation for gastrointestinal endoscopy with sedation. The prospective multicentre randomised controlled ODEPHI study protocol. BMJ Open. 2020 Feb 18;10(2):e034701. doi: 10.1136/bmjopen-2019-034701. PMID 32075842